CLINICAL TRIAL: NCT06509802
Title: Efficacy of an Integrated Growth Mindset Intervention on Reducing Anxiety for Social Work and/or Counselling Practicum Trainees: Study Protocol for a Two-Arm Randomised Controlled Trial
Brief Title: Web-based Single-session Intervention of Mindset for Improving Pre-practicum Anxiety and Coping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20240512001
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Anxiety
Keywords: implicit theory; growth mindset; social work students; counselling students; practicum; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) (Experimental): We-SMILE introduces growth mindsets about intelligence, failure, and negative emotions to pre-practicum trainees, consisting of five components: (a) an introduction to a proactive mindset, including neuroplasticity, the malleability of intelligence and emotion, and the importance of failure and feedback in the learning process; (b) stories and testimonials during practicum which emphasise the belief in change; (c) short videos about allegories of developing intelligence, emotion, and failure mindsets; (d) common questions and misconceptions about growth mindsets; and (e) self-persuasive writing exercises in which participants write down their thoughts and suggestions for others about growth mindsets.
  Interventions: Behavioral: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE)
- Training as usual group (No Intervention): The training-as-usual group will continue the normal training and will be provided with repeated assessments at the same timeframe as the intervention group. Participants in training-as-usual group will receive the intervention course after finishing the eight-week follow-up questionnaire.

INTERVENTIONS:
Behavioral: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) — This study will be a two-arm randomised controlled trial to examine the efficacy of the We-SMILE for pre-practicum social work and/or counselling students by comparing to the We-SMILE intervention group and the no-intervention training-as-usual group.
  Arms: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE)

SUMMARY:
Practicum is an essential educational component of professional training, however, the process can be challenging and sometimes frustrating, with obstacles such as the rigorous training process and mental distress. Being adequately prepared to confront the challenges and difficulties in practicum is crucial for the learning outcomes and psychological well-being of social work and/or counselling trainees. At the same time, mindset is found to be a modifiable factor in intervention, which is essential in clinical psychology, therapy, prevention, and early intervention. Instilling growth mindsets regarding intelligence, emotion, and failure-is-enhancing mindsets, respectively, is worthwhile in easing anxiety and stress coping. However, the existing intervention approaches lack of mindset integration, low intensity, distinctions of employees and interns, more objective and reliable outcome indictors and well-designed randomised controlled trials.

Using a two-arm randomised controlled trial, the proposed study will examine the efficacy of a Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) on reducing anxiety related to practicum and improving mental health and practicum-related outcomes.

A total of 117 students will be recruited from the social work and/or counselling programmes, and randomly assigned to existing pre-practicum training (Training As Usual, TAU) or that plus the We-SMILE. The intervention is 45 minutes in length. Participants will be assessed at three timepoints: baseline (T1), two weeks post-intervention (T2), and eight weeks post-intervention (T3). Patient and public involvement is adopted in the intervention design and implementation strategies. It is expected that the We-SMILE group will present lower anxiety related to practicum and more positive secondary outcomes (depression, anxiety, stress, psychological well-being, learning and performance orientation, academic self-efficacy, and confidence) compared to the TAU group. The intention-to-treat principle and linear-regression-based maximum likelihood multi-level models will be used for data analysis.

The study will not only provide evidence on integrated mindset intervention for trainees' mental health and learning outcomes, but also benefit social work and/or counselling supervisors and programmes as an accessible module.

ELIGIBILITY:
Pre-practicum students in social work and/or counselling programmes are eligible.

* Inclusion Criteria: students who

  1. are about to start the practicum soon;
  2. can read and write Chinese;
  3. consent to participate.
* Exclusion Criteria: students who

  1. do not consent to participate;
  2. cannot concentrate for at least 45 minutes to complete the intervention and questionnaires;
  3. have a disability or serious physical or mental illness resulting in poor condition;
  4. do not participate in the practicum.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety related to practicum | Baseline
  Anxiety related to practicum will be measured by four items, including "level of anxiety about starting the practicum", "how much your anxiety will interfere with their learning", "how prepared you are for the practicum" and "how excited you are to participate in the practicum". Each statement will be rated on a 10-point Likert scale, ranging from 1=completely not anxious, very small, completely unprepared, and completely unexcited to 10=extremely anxious, very great, perfectly prepared, and extremely excited.
Anxiety related to practicum | Two-week post-intervention
  Anxiety related to practicum will be measured by four items, including "level of anxiety about starting the practicum", "how much your anxiety will interfere with their learning", "how prepared you are for the practicum" and "how excited you are to participate in the practicum". Each statement will be rated on a 10-point Likert scale, ranging from 1=completely not anxious, very small, completely unprepared, and completely unexcited to 10=extremely anxious, very great, perfectly prepared, and extremely excited.
Anxiety related to practicum | Eight-week post-intervention
  Anxiety related to practicum will be measured by four items, including "level of anxiety about starting the practicum", "how much your anxiety will interfere with their learning", "how prepared you are for the practicum" and "how excited you are to participate in the practicum". Each statement will be rated on a 10-point Likert scale, ranging from 1=completely not anxious, very small, completely unprepared, and completely unexcited to 10=extremely anxious, very great, perfectly prepared, and extremely excited.

SECONDARY OUTCOMES:
Depression, anxiety and stress | Baseline
  Depression, anxiety, and stress will be assessed by the simplified 12-item Depression Anxiety Stress Scales (DASS-12). The items of DASS-12 were shortlisted from the DASS-21 such as "I found it hard to wind down.". Each item will be rated from 0=never to 4=almost always according to the participant's status over the past week.
Depression, anxiety and stress | Two-week post-intervention
  Depression, anxiety, and stress will be assessed by the simplified 12-item Depression Anxiety Stress Scales (DASS-12). The items of DASS-12 were shortlisted from the DASS-21 such as "I found it hard to wind down.". Each item will be rated from 0=never to 4=almost always according to the participant's status over the past week.
Depression, anxiety and stress | Eight-week post-intervention
  Depression, anxiety, and stress will be assessed by the simplified 12-item Depression Anxiety Stress Scales (DASS-12). The items of DASS-12 were shortlisted from the DASS-21 such as "I found it hard to wind down.". Each item will be rated from 0=never to 4=almost always according to the participant's status over the past week.
Psychological well-being | Baseline
  Psychological well-being will be measured using the seven-item Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). One example item is "I've been feeling optimistic about the future.". Each item is rated from 1 (None of the time) to 5 (All of the time).
Psychological well-being | Two-week post-intervention
  Psychological well-being will be measured using the seven-item Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). One example item is "I've been feeling optimistic about the future.". Each item is rated from 1 (None of the time) to 5 (All of the time).
Psychological well-being | Eight-week post-intervention
  Psychological well-being will be measured using the seven-item Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). One example item is "I've been feeling optimistic about the future.". Each item is rated from 1 (None of the time) to 5 (All of the time).
Learning and performance orientation | Baseline
  Learning and performance orientation will be assessed by eleven adapted items, with five items measuring the learning orientation (e.g., "I like to learn new knowledge in practicums.") and six items measuring performance orientation (e.g., "I like to seek rewards in short term for my efforts."). Each item will be rated by a five-point Likert scale from 1=strongly disagree to 5=strongly agree.
Learning and performance orientation | Two-week post-intervention
  Learning and performance orientation will be assessed by eleven adapted items, with five items measuring the learning orientation (e.g., "I like to learn new knowledge in practicums.") and six items measuring performance orientation (e.g., "I like to seek rewards in short term for my efforts."). Each item will be rated by a five-point Likert scale from 1=strongly disagree to 5=strongly agree.
Learning and performance orientation | Eight-week post-intervention
  Learning and performance orientation will be assessed by eleven adapted items, with five items measuring the learning orientation (e.g., "I like to learn new knowledge in practicums.") and six items measuring performance orientation (e.g., "I like to seek rewards in short term for my efforts."). Each item will be rated by a five-point Likert scale from 1=strongly disagree to 5=strongly agree.
Academic self-efficacy | Baseline
  Academic self-efficacy will be measured by five adapted items. Example items are "I believe that as long as I study diligently, I will be able to master practical skills." and "As long as I am diligent, I can master all of the skills learned during the internship.". The items will be scored from 1=strongly disagree to 5=strongly agree.
Academic self-efficacy | Two-week post-intervention
  Academic self-efficacy will be measured by five adapted items. Example items are "I believe that as long as I study diligently, I will be able to master practical skills." and "As long as I am diligent, I can master all of the skills learned during the internship.". The items will be scored from 1=strongly disagree to 5=strongly agree.
Academic self-efficacy | Eight-week post-intervention
  Academic self-efficacy will be measured by five adapted items. Example items are "I believe that as long as I study diligently, I will be able to master practical skills." and "As long as I am diligent, I can master all of the skills learned during the internship.". The items will be scored from 1=strongly disagree to 5=strongly agree.
Confidence related to practicum | Baseline
  Confidence related to practicum will be assessed by a six-item self-developed scale. Items generated from interviews with social work students, such as "I am confident that I can listen to comments from supervisors/colleagues/service users with an open mind." and "I am confident that I can manage my time well and cope with my practicum work and schoolwork at the same time.". Each item needs to be rated from 1=strongly disagree to 5=strongly agree.
Confidence related to practicum | Two-week post-intervention
  Confidence related to practicum will be assessed by a six-item self-developed scale. Items generated from interviews with social work students, such as "I am confident that I can listen to comments from supervisors/colleagues/service users with an open mind." and "I am confident that I can manage my time well and cope with my practicum work and schoolwork at the same time.". Each item needs to be rated from 1=strongly disagree to 5=strongly agree.
Confidence related to practicum | Eight-week post-intervention
  Confidence related to practicum will be assessed by a six-item self-developed scale. Items generated from interviews with social work students, such as "I am confident that I can listen to comments from supervisors/colleagues/service users with an open mind." and "I am confident that I can manage my time well and cope with my practicum work and schoolwork at the same time.". Each item needs to be rated from 1=strongly disagree to 5=strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Shimin Zhu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Xi A, Wong SSK, Yam K, Leung JTY, Zhu S. Efficacy of a Web-Based Integrated Growth Mindset Intervention on Reducing Anxiety Among Social Work and Counseling Practicum Trainees: Protocol for a 2-Arm Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 27;14:e67234. doi: 10.2196/67234. PMID 40146991